CLINICAL TRIAL: NCT05628194
Title: SAVE THE BOTTOMS!!!: ASSESSING THE GAY MALE EXPERIENCE WITH ANAL CANCER PREVENTION STRATEGIES
Brief Title: ASSESSING THE GAY MALE EXPERIENCE WITH ANAL CANCER PREVENTION STRATEGIES
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: HRP-580
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Anal Cancer
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Men who have sex with men (MSM)
  Interventions: Other: Observational/Survery

INTERVENTIONS:
Other: Observational/Survery — MSM participants will complete a one-time survey, delivered in an e-format. Survey will be accessible via Meta-based social media platforms (Facebook, Instagram).

SUMMARY:
The purpose of this study is to describe current knowledge and opinions about anal cancer screening among men who have sex with men (MSM), as well as their experience receiving guideline-compliant care aimed at anal cancer risk reduction using a large-scale survey disseminated via social media.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Current resident of the U.S.
* Engage in anoreceptive intercourse with male partners
* Fluent in English or Spanish

Exclusion Criteria:

* Under the age of 18 years old
* Not living in the United States
* Not born with sex assigned at birth as male
* Does not engage in sex with male partners

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: MSM population, which may include individuals who may identify as having a sexual orientation of gay, bisexual, or gender-queer. They may identify as any gender, including trans-gender or non-binary (but limited to those born with sex assigned at birth as male).
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
MSM awareness of anal cancer risk | 2 months
  Survey with question items on participants' awareness of anal cancer risk
MSM awareness of strategies to decrease anal cancer risk | 2 months
  Survey with question items of strategies to decrease anal cancer risk

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Arsoniadis, M.D., Ph.D, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No